CLINICAL TRIAL: NCT05153681
Title: Comparison of Peloid Therapy and Kinesio Tape Effectiveness in Patients With Plantar Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Süleyman Gül, Physician, Konya Meram State Hospital
Other Study IDs: KonyaMeramSH
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Plantar Fasciitis
Keywords: mud therapy; balneotherapy; athletic Tape
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Mud Therapy; Athletic Tape

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peloid Therapy: Peloidotherapy is a special balneotherapy method made with natural mud. In both domestic and international scientific studies on peloid treatment, it has been shown that pain in patients decreases, physical functions improve, quality of life increases, and the amount of painkillers use decreases.
  Interventions: Other: Peloid Therapy
- Kinesio Tape: Kinesio tapes, which have been used in the conservative treatment of plantar fasciitis in recent years, are elastic tapes similar to the structural properties and flexibility of human skin, without limiting joint movements.
- Home exercise: In addition to the cold application, gastrocnemius and plantar fascia stretching and strengthening exercises were applied to patients with plantar fasciitis.

INTERVENTIONS:
Other: Peloid Therapy — Peloid therapy; A total of 10 sessions were applied for 30 minutes by heating the proximal part of the sole of the foot, including the heel part, at a temperature of 45 degrees. Kinesioband application: One strip is prepared as a rake with a length of about 25 cm, and the other strip is prepared as an I tape with a length of about 20 cm. The ankle is in a neutral position of 90 degrees. Lymphatic and mechanical correction technique is applied. Afterwards, the band is activated.
  Other Names: Home exercise; Kinesio tape
  Groups: Peloid Therapy

SUMMARY:
The Plantar Fascia (PF) is a thick, fibrous sheath located in the middle of the sole of the foot, starting from the tuber calcanei in the calcaneus and extending to the level of the middle phalanges. Plantar Fasciitis (PFs) is inflammation and thickening of the PF where it attaches to the calcaneus. PFs are the most common cause of heel pain. Diagnosis is made by physical examination and radiological examinations. On physical examination, there is localized tenderness medial to the calcaneal tuberosity. In the treatment of plantar fasciitis, there are many applied methods such as anti-inflammatory agents, orthostotic supports, night splints, physical therapy, corticosteroid applications, night splint use, plastering, rest, lifestyle modification, laser, taping, exercise and ESWT. Kinesio tapes, which have been used in the conservative treatment of plantar fasciitis in recent years, are elastic tapes similar to the structural properties and flexibility of human skin, without limiting joint movements. Peloidotherapy is a special balneotherapy method made with natural mud. In both domestic and international scientific studies on peloid treatment, it has been shown that pain in patients decreases, physical functions improve, quality of life increases, and the amount of painkillers use decreases. We could not find any study comparing Peloidotherapy and Kinesioband methods routinely used in the treatment of PF in the literature.

DETAILED DESCRIPTION:
The Plantar Fascia (PF) is a thick, fibrous sheath located in the middle of the sole of the foot, starting from the tuber calcanei in the calcaneus and extending to the level of the middle phalanges. It is a tendinous aponeurosis rather than a true layer of fascia and is an important static support for the longitudinal arch of the foot. Plantar Fasciitis (PFs) is inflammation and thickening of the PF where it attaches to the calcaneus. PFs are the most common cause of heel pain. It has been reported to occur in 10% of people during their lifetime. It is more common between the ages of 40-60. Although its main etiology is not fully understood, the most common theory is; microscopic tears as a result of mechanical overstretching of the fascia followed by chronic inflammation, but histological studies lack evidence to support inflammation. Diagnosis is made by physical examination and radiological examinations (ultrasonography, radiography). On physical examination, there is localized tenderness medial to the calcaneal tuberosity. In the treatment of plantar fasciitis, there are many applied methods such as anti-inflammatory agents, orthostotic supports, night splints, physical therapy, corticosteroid applications, night splint use, plastering, rest, lifestyle modification, laser, taping, exercise and ESWT.

Kinesio tapes, which have been used in the conservative treatment of plantar fasciitis in recent years, are elastic tapes similar to the structural properties and flexibility of human skin, without limiting joint movements. Kinesio taping technique provides physiological effects on skin, fascia, muscle and joint. After applying kinesio tape, it raises the skin in the taped area, increasing the space between it and the muscles and relieving the pressure in that area. It also helps to reduce tension and sensitivity by increasing blood circulation and prevents stimulation of pain receptors.

Peloids (medical mud) are organic or inorganic substances formed as a result of geological and/or biological events. They can be found in nature as fine particles, or they are made into small, fine particles by some preliminary preparation processes. Peloidotherapy is a special balneotherapy method made with natural mud. It is used in the treatment of diseases such as degenerative joint diseases, soft tissue rheumatism, lumbardiscopathy, cervical discopathy, chronic low back and neck pain, joint pain. In both national and international scientific studies on peloid treatment, it has been shown that pain in patients decreases, physical functions improve, quality of life increases, and the amount of painkillers use decreases.

We could not find any study comparing Peloidotherapy and Kinesioband methods routinely used in the treatment of PF in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Pain on the sole of the foot for six weeks or longer,
* Being between the ages of 18-65,
* Pain that is 4 or more severe according to VAS,
* Localized tenderness on palpation medial to the calcaneal tuberosity,
* Heel pain when getting out of bed in the morning or after long periods of inactivity

Exclusion Criteria:

* Having neuropathic or radicular pain,
* Acute ankle trauma,
* Having surgical intervention on the heel before,
* Receiving non-operative treatment for the heel and sole in the last 6 months (corticosteroid injection, physical therapy applications, ESWT etc.),
* Presence of rheumatological diseases such as rheumatoid arthritis, psoriatic arthritis,
* Having orthopedic deformity in the foot/ankle,
* Those with a history of uncontrollable systemic disease (cardiovascular, pulmonary, hepatic, renal, hematological..),
* Those with a history of systemic endocrine disease (DM, hyperthyroidism..),
* History of major psychiatric illness
* Bleeding disorders and those using anticoagulants
* Those with malignancy,
* Being allergic to peloid therapy,
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 105 patients, 35 for peloid treatment, 35 for Kinesio tape, and 35 for home exercise, were included in our study.
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficacy of kinesio tape and peloid therapy in patients with plantar fasciitis | October 2020-February 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No